CLINICAL TRIAL: NCT04918329
Title: Observatory of Functionnal Digestive Disorders
Brief Title: Functional Digestive Disorders Observatory
Acronym: OTFI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Anne Marie LEROI, Principal Investigator, University Hospital, Rouen
Other Study IDs: 2019/120/OB; 2019/120/OB (Registry Identifier: Functional Digestive Disorders Observatory)
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia; Functional Constipation; Faecal Incontinence; Abdominal Pain (AP); Vomiting Syndrome
Keywords: Observatory; functional digestive disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia; Encopresis; Abdominal Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, fecaes, biopsies, urine,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Non interventional study
  Other Names: Non interventional study

SUMMARY:
Functional digestive pathologies are defined by symptoms such as functional dyspepsia, gastroesophageal reflux, irritable bowel syndrome, gastroesophageal reflux, functional constipation, functional diarrhea, functional bloating, the opioid-induced constipation and fecal incontinence, without organic substratum. These diseases are very common in the general population (20%) and represent the first cause of consultation in city gastroenterology. The pathophysiology of these functional disorders is complex and often multifactorial: disturbances in digestive motility, altered visceral sensitivity, sphincter dysfunction, post-surgery, intestinal inflammation, dysbiosis, and impairment of the gut-brain axis. For example, it has been shown that one in four patients with inflammatory bowel disease in confirmed remission report digestive symptoms consistent with a functional bowel disorder, suggesting a possible pathophysiological continuum between these two conditions.

The objective of this study is to collect prospective clinical and tests data and a biological collection from biological samples (digestive biopsies, blood, urine and fecal samples) collected as part of the standard care. This collection could identify diagnostic or prognostic markers of the therapeutic response.

DETAILED DESCRIPTION:
Functional digestive pathologies are defined by symptoms such as functional dyspepsia, gastroesophageal reflux, irritable bowel syndrome, gastroesophageal reflux, functional constipation, functional diarrhea, functional bloating, the opioid-induced constipation and fecal incontinence, without organic substratum. These diseases are very common in the general population (20%) and represent the first cause of consultation in city gastroenterology.

The pathophysiology of these functional disorders is complex and often multifactorial: digestive motility disorders, digestive sensitivity disorders, sphincter dysfunction, post-surgery, intestinal inflammation, dysbiosis, disruption of the gut-brain axis. For example, it has been shown that one in four patients with proven remission of chronic inflammatory bowel disease reports digestive symptoms compatible with a functional intestinal disorder, suggesting a pathophysiological continuum between these two conditions.

In our center, patients with functional digestive disorders undergo a comprehensive assessment that evolves in line with scientific advances and the emergence of new diagnostic or prognostic tools. This assessment helps to identify the pathophysiological mechanisms involved in the functional digestive disorder: disturbances in digestive motility, visceral hypersensitivity, mucosal alterations, sub-inflammatory syndrome, and dysfunction of the gut-brain axis. All of these abnormalities may be promoted by a genetic predisposition leading to alterations in neurotransmitters, immune function, mucosal integrity, and so on.

Our objective is to study the pathophysiological mechanisms, including genetic factors, responsible for functional digestive disorders as a whole, whether or not they are sequelae of an organic pathology.

To do that, we collect prospective clinical and tests data and we perform a biological collection from biological samples (digestive biopsies, blood, urine and fecal samples) collected as part of the standard care. This collection could identify diagnostic or prognostic markers of the therapeutic response. The investigators hope that a better knowledge of the pathophysiology of digestive functional diseases will improve the therapeutic management by making a therapeutic choice based on the observed pathophysiological abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patients with functional digestive disorder for more of 3 months;
* Patients assessed as part of routine care;
* Patients affiliated to the Social Security ;
* Patients not opposed to participation in the Centre

Exclusion Criteria:

* Person deprived of liberty by administrative or judicial decision or major protected subject (under guardianship or curatorship);
* Patients unable for any reason to read, understand, respond questionnaires (visual, psychiatric, cognitive, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with functional digestive disorders consulting in our centre functional digestive disorders whether or not they are sequelae of an organic pathology.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2030-10-09 (Estimated); Study Completion 2030-10-09 (Estimated)

PRIMARY OUTCOMES:
Functional digestive explorations | 10 years
  Gastrointestinal intraluminal pressures (mmHg), recorded during gastrointestinal manometry.

SECONDARY OUTCOMES:
Radiological findings | 10 years
  Luminal dimensions (cm)
Clinical data of patients with functional digestive disorders | 10 years
  ethnicity (categorical measure)
Gastric emptying study | 10 years
  Gastric emptying time (minutes)
EndoFLIP system | 10 years
  Cross-sectional area (CSA) (mm²) measured using the EndoFLIP® system.
Rectal barostat | 10 years
  Rectal distension compliance (Ml/mmHg) measured using a rectal barostat.
Breath tests | 10 years
  Percentage of hydrogen (H₂) and methane (CH₄) in exhaled breath during breath testing.
Endoscopic findings | 10 years
  Mucosal abnormalities (caterogical variable)
Drug use | 10 years
  Drug use (categorical variable)
Gastrointestinal symptoms | 10 years
  Rome questionnaire
Gastrointestinal symptoms | 10 years
  Bristol Scale
Gastrointestinal symptoms | 10 years
  Francis score
Gastrointestinal symptoms | 10 years
  GIQLI score
Gastrointestinal symptoms | 10 years
  Cleveland Clinic Score
Gastrointestinal symptoms | 10 years
  FIQL score
Symptoms of anxiety and depression | 10 years
  HAD questionnaire
Sleep assessment | 10 years
  Pittsburgh Sleep Quality Index (PSQI)
Sleep assessment | 10 years
  Insomnia severity index
painful bladder symptom | 10 years
  Painful bladder score
Gastrointestinal symptoms | 10 years
  PAGI-SYM score
Gastrointestinal symptoms | 10 years
  PAGI-QOL
Gastrointestinal symptoms | 10 years
  Reflux questionnaire RDQ
Anxiety and depression syndrome | 10 years
  Patient health questionnaire
Anxiety symptoms | 10 years
  Generalized Anxiety Disorder questionnaire
Gastrointestinal symptoms | 10 years
  Kess score
Anxiety symptoms | 10 years
  Generalized Anxiety Disorder
Gastrointestinal symptoms | 10 years
  Visceral Sensitivity Index (VSI)
Eating behavior assessment | 10 years
  SCOFF questionnaire
Eating behavior assessment | 10 years
  ARFID questionnaire
Sleep assessment | 10 years
  Ford Insomnia Response to Stress Test (FIRST)
Global health assessment | 10 years
  PROMIS 10 Score
Gastrointestinal symptoms | 10 years
  IBSQOL score
General Health Questionnaire | 10 years
  WRQ score
Gastrointestinal symptoms | 10 years
  Gastroparesis questionnaire
Gastrointestinal symptoms | 10 years
  Vaizey questionnaire
Gastrointestinal symptoms | 10 years
  CISS score
Health assessment | 10 years
  EQ-5D-5L
Eating behavior assessment | 10 years
  Fear of food score
Eating behavior assessment | 10 years
  Food avoidance score
Eating behavior assessment | 10 years
  FITAS score
Gastrointestinal symptoms | 10 years
  PAC-QOL
Gastrointestinal symptoms | 10 years
  NBD score
Gastrointestinal symptoms | 10 years
  LARS score
Demographic data | 10 years
  age (years)
Demographic data | 10 years
  sex (categorical measure)
Gastrointestinal treatments | 10 years
  Treatments (categorical measure)

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology Unit, Hopital Charles Nicolle, 1 rue de Germont, Rouen, France

IPD SHARING:
Plan to Share IPD: No
No sharing plan

REFERENCES:
- [Derived] Soliman H, Wuestenberghs F, Desprez C, Leroi AM, Melchior C, Gourcerol G. Physiological characterization of gastric emptying using high-resolution antropyloroduodenal manometry. Am J Physiol Gastrointest Liver Physiol. 2024 Jan 1;326(1):G16-G24. doi: 10.1152/ajpgi.00101.2023. Epub 2023 Oct 24. PMID 37874655
- [Derived] Gourcerol G, Melchior C, Wuestenberghs F, Desprez C, Prevost G, Grosjean J, Leroi AM, Tavolacci MP. Delayed gastric emptying as an independent predictor of mortality in gastroparesis. Aliment Pharmacol Ther. 2022 Apr;55(7):867-875. doi: 10.1111/apt.16827. Epub 2022 Feb 20. PMID 35187671